CLINICAL TRIAL: NCT04330248
Title: An Open-label, Single-sequence, Drug-drug Interaction Study to Evaluate the Effect of Steady-state Carbamazepine on the Single-dose Pharmacokinetics of Erdafitinib Tablets in Healthy Adult Subjects
Brief Title: A Study of Steady-state Carbamazepine on the Single-dose of Erdafitinib Tablets in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108763; 2019-003473-26 (EudraCT Number); 42756493NAP1001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — erdafitinib; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erdafitinib and Carbamazepine (Experimental): Participants will receive single oral dose of erdafitinib dose 1 on Day 1 30 minutes after the start of a standardized breakfast in Period 1 followed by repeated doses of carbamazepine orally every 12 hours from Days 15 to 35 (carbamazepine Dose 1 from Days 15 to 17, Dose 2 from Days 18 to 20, and then Dose 3 from Days 21 to 35) 30 minutes after the start of standardized meal (breakfast and dinner) in Period 2. After 8 Days of Dose 3 carbamazepine treatment, on Day 28, participants will receive a single oral dose of erdafitinib dose 1 with that day's carbamazepine dose.
  Interventions: Drug: Erdafitinib; Drug: Carbamazepine

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive single oral dose of erdafitinib tablets on Day 1 in Period 1 and on Day 28 in Period 2.
  Other Names: JNJ-42756493
Drug: Carbamazepine — Participants will receive an oral dose of carbamazepine tablets from Day 15 to 35 in Period 2.

SUMMARY:
The main purpose of this study is to evaluate the effect of multiple doses of carbamazepine (a strong inducer of cytochrome P450 [CYP]3A4 and a weak inducer of CYP2C9) on the pharmacokinetics of a single oral dose of erdafitinib in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs (blood pressure, pulse, and body temperature) performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel and hematology panel are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator. Participants must have sodium and phosphate levels within normal limits; hematological parameters (Hemoglobin, red blood cell [RBC] count, white blood cell [WBC] count, absolute neutrophil count, platelet count) within normal limits; and total bilirubin, alanine aminotransferase (ALT), aspartate amino transferase (AST), and alkaline phosphatase (ALP) serum levels lower than or equal to the upper limit of normal at screening
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Must agree to have a pharmacogenomic blood sample (5 milliliters [mL]) collected at screening to allow for pharmacogenomic analysis
* Non-smoker for at least 6 months before first study drug administration

Exclusion Criteria:

* History of depression or suicidal ideation
* History or current evidence of ophthalmic disorder, such as central serous retinopathy (CSR) or retinal vein occlusion, active wet age-related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation, or ulceration
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (a maximum of 3 doses per day of 500 milligram [mg] paracetamol, and no more than 3 gram [g] per week), hormonal replacement therapy and cetirizine (in case of allergic reactions), within 14 days before the first dose of the study drug is scheduled until completion of the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 5 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Known allergies, hypersensitivity, or intolerance to erdafitinib or carbamazepine or any of the excipients of the formulations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma (Cmax) of Erdafitinib | Predose (Day 28) 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168 and 312 hours postdose (Day 41)
  Cmax is defined as the maximum observed plasma of erdafitinib concentration.
Area Under the Plasma Analyte Concentration-Time Curve 0 from Time 0 to one week Postdose (AUC[0-168 hours]) | Predose (Day 28) 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose (Day 35)
  AUC (0-168 hours) is defined as the area under the plasma analyte concentration-time curve from time 0 to one week postdose (168 hours).
Area Under the Plasma Analyte Concentration-Time Curve from Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) | Predose (Day 28) 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168 and 312 hours postdose (Day 41)
  AUC (0-last) is defined as area under the plasma analyte concentration-time curve from time 0 to time of the last observed quantifiable concentration.
Area Under the Analyte Concentration-Time Curve from Time 0 to Infinite Time (AUC [0-infinity]) | Predose (Day 28) 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168 and 312 hours postdose (Day 41)
  AUC (0-infinity) is defined as the area under the analyte concentration-time curve from time 0 to infinite time.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Day 79 (end of study)
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency